CLINICAL TRIAL: NCT04434313
Title: Treatment of Hemiparetic Gait Impairments Using Telehealth With the Moterum iStride Solution™
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Moterum Technologies, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MOT-TELE-2020-04-00
Record Dates: First submitted 2020-06-03; First posted 2020-06-16 (Actual); Last update posted 2022-09-07 (Actual); Status verified 2022-09

CONDITIONS: Telemedicine; Gait, Hemiplegic; Gait Disorders, Neurologic; Stroke; Orthotic Devices; Gait Analysis
Keywords: iStride; Telehealth; Telerehabilitation; Gait Speed
MeSH Terms: conditions — Gait Disorders, Neurologic; Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Delivery of iStride™ device gait treatment using telemedicine (Experimental): Treatment with the gait device will be adapted to remote delivery using the telemedicine platform. Participants and caregivers will be guided through an adapted treatment protocol remotely by physical therapists. Training will include platform navigation, device instruction, treatment guidelines, safety precautions, and assessment performance. Understanding will be verified through a caregiver quiz.
  Gait patterns will be monitored before, during, and after treatment using gait sensors and outcome measures. Assessments include the 10-Meter Walk Test, Six Minute Walk Test, Timed Up and Go Test, Geriatric Depression Scale, Activities-Specific Balance Confidence Scale, and Stroke Impact Scale-16. Treatment will consist of 12 sessions of walking on the device for a goal of 30 minutes per session. Assessments will be repeated one-week, one-month, three-months, six-months, and 12-months after treatment. Feasibility and safety of the delivery method will be measured throughout the trial.
  Interventions: Device: Delivery of iStride™ device gait treatment using telemedicine

INTERVENTIONS:
Device: Delivery of iStride™ device gait treatment using telemedicine — The gait device used in this study mimics the actions of the split-belt treadmill but can be used during overground walking and in one's own home, thus enabling long-term training. This device does not require any external power and is completely passive; all necessary forces are redirected from the natural forces present during walking. This research aims to adapt the delivery mechanism of treatment with the iStride™ device to include telemedicine. The telemedicine platform of reference in this study, the Moterum Digital Platform, is an integrated therapeutic platform which offers an activity library, real-time video conferencing, and outcomes tracking. Our primary study objective is to determine if telemedicine is a safe and feasible delivery method for treatment with the iStride ™ gait device.

SUMMARY:
The objective of this research is to investigate the feasibility of delivering gait treatment using the Moterum iStride Solution™ to individuals with hemiparetic gait impairments using a telemedicine modality, the Moterum Digital Platform.

DETAILED DESCRIPTION:
Hemiparesis, a common disabling consequence of stroke and other neurologic conditions, can lead to abnormal gait function often characterized by asymmetric patterns and decreased gait speed. A large percentage of stroke survivors, up to 70%, experience gait dysfunction, which can lead to reduced activity levels, limited community participation, and contribute to an increased risk of falls. Effective interventions to treat gait dysfunction are essential to reduce disability for these individuals.

The iStride™ gait device, initially designed to mimic the symmetry-improving mechanism of a split-belt treadmill, was developed to treat asymmetric gait impairments in stroke survivors. Unlike many currently available gait treatment devices, the iStride™ device is portable, therefore allowing gait treatment to occur overground and from the home environment. Training in natural environments is believed to enhance the transfer of learning as well as enable long-term training. Previously published studies with the iStride™ device demonstrate its ability to beneficially improve functional gait parameters, gait speed, and reduce fall risk in both clinical and home settings.

To monitor improvement in gait function, the device is paired with patented iStride sensors™. The combined system, the Moterum iStride Solution™, is currently being used by stroke survivors in the home environment. In the current delivery model, users are provided instruction and training from physical therapists in clinical settings before using the device in their home environment under the supervision of a Moterum staff member. User feedback has led to the exploration of novel methods to deliver device treatment remotely. [Additionally, the need for remote treatment has increased in urgency with the onset of the coronavirus pandemic and social distancing guidelines.]

In this study, treatment with the iStride™ will be adapted to remote delivery using a telemedicine platform, the Moterum Digital Platform. A screening process will be implemented to guide participant selection and identify individuals likely to be successful with remote treatment delivery using the telemedicine modality. This process consists of an initial eligibility criteria review followed by a physical therapist video review of participant walking patterns.

Once enrolled in the clinical trial, participants will receive study-related equipment including the iStride™ device, Moterum iStride Hub and Sensors™, and a pre-measured strap for gait testing. They will be instructed in the download of the Moterum Digital Platform which will serve as the telemedicine modality for subsequent communication. Participants and their caregivers will be provided with instructional videos as well as therapist training on study procedures using video calls through the telemedicine platform. Instruction will include telemedicine portal navigation, iStride™ fitting (donning/doffing), mobility and walking guidelines with iStride™ device, assessment performance, environmental considerations, safety precautions, and caregiver guidelines and responsibilities.

Changes to gait patterns will be assessed using specialized gait sensors and functional outcome measures before, during, and after the treatment. Caregivers will be trained in the performance of these outcome measures which can be overseen by physical therapists through video conferencing.

Feasibility, compliance, and safety of the delivery method will be investigated throughout the trial using prompted questions within the Moterum Digital Platform and integrated forms to be completed by the participant and/or caregiver. After treatment is completed, participants and their caregivers will be surveyed to obtain feedback regarding usability, satisfaction, and sentiments regarding the remote delivery model.

ELIGIBILITY:
Inclusion Criteria:

* Age 21-80
* Caregiver support. The caregiver should be an adult over the age of 18 without physical or cognitive limitations which would prohibit them from being able to provide appropriate assistance to the device user
* Hemiparesis
* If hemiparesis is due to a stroke, the stroke occurred at least 3 months prior to enrollment
* Gait asymmetry
* Able to walk independently with or without a cane or hemiwalker, (Modified Rankin Score 3 or less)
* No evidence of severe cognitive impairment that would interfere with understanding the instructions
* At least 25 feet of walking space (does not need to be a straight line)
* Weight does not exceed 275lbs

Exclusion Criteria:

* Uncontrolled seizures
* Metal implants (stents, clips, pacemaker)
* Pregnancy
* Chronic Obstructive Pulmonary Disease
* Uncontrolled blood pressure
* Myocardial infarction within the last 180 days
* Cannot rely on a rolling walker for ambulation
* Severe ataxia interfering with safety on the device
* Previously diagnosed vestibular ear issues interfering with safety on the device

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2020-04-20 (Actual); Primary Completion 2020-12-19 (Actual); Study Completion 2020-12-21 (Actual)

PRIMARY OUTCOMES:
Feasibility of safely implementing the treatment protocol | Determined at the end of the 12-session treatment period (approximately 4 weeks after beginning the treatment).
  The described delivery method includes using remote physical therapist treatment oversight and physical supervision of treatment activities by trained caregivers. Due to the inclusion criteria, patients already have some risk of falls and need for assistance while walking. The caregivers will record assistance levels provided during treatment. Any adverse events will be immediately reported and reviewed. The remote physical therapists will regularly review assistance levels to ensure the participant is requiring an appropriate level of assistance. The feasibility of safely delivering treatment will be assessed by two measures: (a) the daily safety rate, defined as the percentage of days an adverse event occurred out of the total number of treatment days, and (2) assistance required and adverse events experienced for each participant, compared to the group, and compared to our prior research.
Achievability of telemedicine delivery protocol | Determined within one week after the final follow-up assessment (12-month follow-up) is completed. The 12-month follow-up assessment will occur 12-months after completion of the 4-week treatment period.
  The achievability of this treatment delivery method will be assessed by measuring participant compliance to the protocol tasks. These tasks include scheduled treatment sessions, functional and psychosocial outcome measures, and sensor-based activities. Achievability will be defined as the percentage of completed protocol activities out of the total scheduled activities.

SECONDARY OUTCOMES:
Feasibility of screening criteria | Determined at the end of the 12-session treatment period (approximately 4 weeks after beginning the treatment).
  To enroll patients via telemedicine, the eligibility criteria will be assessed with an additional video gait review performed by physical therapists. The feasibility of screening patients at a distance will be assessed by measuring screening performance, defined as the percentage of enrolled subjects who are removed from the study after later being deemed ineligible (for example, gait is not asymmetric or hemiparetic but appeared so on video, or patient cannot walk independently, etc.) out of all enrolled subjects.
Stakeholder Acceptability | Determined within one week after the final follow-up assessment (12-month follow-up) is completed. The 12-month follow-up assessment will occur 12-months after completion of the 4-week treatment period.
  Participant and caregiver feedback will be necessary to determine preferences and sentiments regarding the delivery method including technology management, training procedures, protocol activities, adequacy of caregiver and therapist support, device benefit, and overall satisfaction with procedures. Feedback will be gathered through a questionnaire using five-point Likert scales and open-ended questions. Questionnaires will be provided after completion of outcome measures at the final, 12-month follow-up assessment. Acceptability will be determined through percentage of positive responses out of the total questionnaire items.

CONTACTS AND LOCATIONS:
Overall Officials: Stephen T. Shultz, PT, DPT, OCS, Principal Investigator — Wingate University
Locations (1):
- Moterum Technologies, Inc. (study location: homes throughout United States), Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Reed KB, Handzic, Ismet, Inventor; University of South Florida, assignee. Gait Altering Shoes. US patent 9,295,302. March 29, 2016, 2016.
- [Background] Handzic I, Vasudevan E, Reed KB. Developing a Gait Enhancing Mobile Shoe to Alter Over-Ground Walking Coordination. IEEE Int Conf Robot Autom. 2012 May;2012:4124-4129. doi: 10.1109/ICRA.2012.6225346. PMID 23484067
- [Background] Handzic I, Barno EM, Vasudevan EV, Reed KB. Design and Pilot Study of a Gait Enhancing Mobile Shoe. Paladyn. 2011 Dec 1;2(4):10.2478/s13230-012-0010-7. doi: 10.2478/s13230-012-0010-7. PMID 24371521
- [Background] Kim SH, Huizenga DE, Handzic I, Ditwiler RE, Lazinski M, Ramakrishnan T, Bozeman A, Rose DZ, Reed KB. Relearning functional and symmetric walking after stroke using a wearable device: a feasibility study. J Neuroeng Rehabil. 2019 Aug 28;16(1):106. doi: 10.1186/s12984-019-0569-x. PMID 31455358
- [Derived] Darcy B, Rashford L, Shultz ST, Tsai NT, Huizenga D, Reed KB, Bamberg SJM. Gait Device Treatment Using Telehealth for Individuals With Stroke During the COVID-19 Pandemic: Nonrandomized Pilot Feasibility Study. JMIR Form Res. 2023 May 19;7:e43008. doi: 10.2196/43008. PMID 37204830